CLINICAL TRIAL: NCT03222726
Title: Chief of Nephrology, Professor, Shanghai Pudong Hospital,
Brief Title: The Study of the Internet Monitoring and Analysis of Exercise to Reduce the Complications of Diabetic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Principal Investigator, Jin HM, MD, Professor, Shanghai Pudong Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ShanghaiPudongH
Record Dates: First submitted 2017-07-18; First posted 2017-07-19 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-04

CONDITIONS: Exercise
Keywords: exercise, diabetic kidney disease, complications
MeSH Terms: conditions — Motor Activity; Diabetic Nephropathies

STUDY DESIGN:
Intervention Model Description: corhort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Active Comparator): 6000 steps/day or 40,000 steps/week
  Interventions: Other: exercise group
- less-exercise group (Other): less than 6000 steps/day or 40,000 steps/week
  Interventions: Other: exercise group

INTERVENTIONS:
Other: exercise group — less than 6000 steps/day or 40,000 steps/week
  Other Names: less-exercise group

SUMMARY:
Microvascular complications are a major complication of diabetes.Diabetic microvascular complications can not only lead to chronic kidney disease and retinopathy, but also affect the quality of life of patients with diabetic nephropathy, which can lead to the death of diabetic patients.Due to diabetes patient survival for decades, in spite of more than 90% of time is a life outside the hospital, so the analysis of the effect of outside risk factors for complications of hospital and progress, and to find effective intervention measures is of great significance for the prevention and control of diabetic microvascular complications.Therefore, we use of advanced Internet technology, and analysis of large data algorithms, and try to keep track of routine indicators such as the patient's urine in real time in patients' families.

This topic mainly observe movement (step 6000 steps per day or 6000 / week) in patients with type 2 diabetic kidney disease microvascular end point events, provide the basis for prevention and control of diabetes kidney complications, clinical significance and treatment prospects.

DETAILED DESCRIPTION:
Research target:To explore exercise intervention in patients with diabetic nephropathy (intervention time for 3 years), the events in the primary end point was observed (double serum creatinine, ESRD dialysis) and secondary events (reduced urinary protein and retinopathy progression, cardiovascular events, and cerebrovascular events for all-cause mortality).

Major technical programmes:

The research object:Clinical diagnosis of type 2 diabetic nephropathy patients. The inclusion criteria: Clinical diagnosis of type 2 diabetic nephropathy patients.Many years history of diabetes, urinary albumin excretion rate of more than 30-300 mg/L, eye exams have diabetic retinopathy, routine urine without red blood cells, double renal morphologic examination being normal, and excludes the other secondary kidney disease. Age 18-75. Willing to participate in this test.

Exclusion criteria: Type 1 diabetes, with other systemic diseases such as cancer, liver function damage, severe edema, cardiac insufficiency (grade 3, 4, cardiac function disorder), serious lung disease caused by respiratory insufficiency, pregnancy and lactation women, and could not walk and did not sign the informed consent of the patients.

Estimate the sample size: In this study, the incidence of the combined endpoint was 40% in the untreated group, 30% in the treatment group, 10% in the treatment group and 80% in the control group, and 0.05 in bilateral statistical level. The above formulations are calculated by each group of 112 cases; Therefore, the sample size of this study is 120 cases per group.

Corhort study: Exercise group (walking 6000 steps or more than 40,000 steps on foot), non-exercise group (walking 6000 steps or less than 40,000 steps on foot).

Follow-up examization: Check the routine of morning urine daily, and check the blood sugar, HbA1c, fasting insulin level, kidney function, liver function, electrolyte, blood routine, blood c-reactive protein and blood type B natriuretic peptide per quarter.

Kidney endpoint event: The blood creatinine was doubled on baseline, or the eGFR was assessed for end-stage renal disease and required dialysis or transplantation.

Cardiovascular endpoint event: During the observation, cardiac failure and acute myocardial infarction were defined as cardiac endpoints Cerebrovascular endpoint event: Hospitalization of cerebral stroke or cerebral hemorrhage is defined as the end of the brain.

Retinal progression: The severity of retinopathy was analyzed based on the fundus photographs, according to Early Treatment Diabetic Retinopathy Study (ETDRS)(1. Benefits of Renin-Angiotensin Blockade on Retinopathy in Type 1 Diabetes Vary With Glycemic Control. Diabetes Care 2011; 34:1838-1842。2. Renal and Retinal Effects of Enalapril and Losartan in Type 1 Diabetes. N Eng J Med 2009; 361:40-51).

Adverse reactions: The adverse reactions of the movement include collapse, body weakness and muscle soreness are recorded.

Internet web system: The urine is monitored outside the general hospital, and The patient urine routine test results were tracked in real time by the external follow-up system of subekang internet web system.

Monitor steps:Add patients' buddy feature to WeChat to add the WeChat movement public number to see the number of steps on the WeChat public number.

ELIGIBILITY:
Inclusion Criteria: Patients with type 2 diabetic nephropathy were diagnosed clinically. Diagnostic criteria: there are many years of history of diabetes, urinary albumin excretion rate of more than 30-300 mg/L, eye exams have diabetic retinopathy, routine urine without red blood cells, double renal morphologic examination is normal (no obstruction after kidney), and excludes the other secondary kidney disease. Age 18-75. Willing to participate in this test.

-

Exclusion Criteria: Type 1 diabetes, with other systemic diseases such as cancer, liver function damage, severe edema, cardiac insufficiency (grade 3, 4, cardiac function disorder), serious lung disease caused by respiratory insufficiency, pregnancy and lactation women, and could not walk and did not sign the informed consent of the patients.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-04-06 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
kidney endpoint | 3-year
  Blood creatinine doubled on baseline, or was evaluated by eGFR and needed for dialysis or transplantation

SECONDARY OUTCOMES:
cardiovascular endpoint | 3-year
  Cardiac failure and acute myocardial infarction were defined as cardiac endpoints
cerebrovascular endpoint | 3 years
  stroke or Cerebral hemorrhage
Retinal progression | 3 years
  The severity of retinopathy was analyzed based on the fundus photographs

CONTACTS AND LOCATIONS:
Overall Officials: Bo Yu, Study Director — Hospital
Locations (1):
- Shanghai Pudong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
study is completed.all data is open in clinicaltrials.gov
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: data will become available when paper published in English journal, and for 5 years